CLINICAL TRIAL: NCT07115498
Title: Piloting a Mobile Adherence Game With Economic Incentives for Young People With HIV in Ghana
Brief Title: Piloting the Incentivized Text-Based Adherence Game Intervention.
Acronym: iTAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Providence College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-FY24-62
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: HIV Treatment Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iTAG (Experimental): Participants in this arm receive the iTAG intervention.
  Interventions: Behavioral: iTAG

INTERVENTIONS:
Behavioral: iTAG — Participants in this intervention start by receiving a brief (15 minute) in-person standard-of-care counseling session focused on increasing their knowledge of HIV treatment adherence and strategies to improve adherence. Following this session, they will then receive daily or less frequent text messages (SMS) over the course of three months. Messages are primary two-way, automated, and have preprogrammed response options. Message content includes HIV medication reminders, motivational messages, information on topics relevant to HIV treatment (e.g., HIV disclosure) in the form of quizzes, opportunities to reach out for support from clinic staff or peer mentors, and game-based messages including story messages, a weekly scoreboard, point system progress, and peer interactions.

SUMMARY:
This project will develop and test a novel intervention to improve HIV treatment adherence among young adults with HIV who attend an HIV clinic in Kumasi, Ghana. The intervention is called incentivized Text-Based Adherence Game (iTAG). It is delivered solely via text messages and includes many advanced features including a point system that rewards participants for responding to texts, a scoreboard that compares participants' progress with each other, and messages on a range of health and HIV-related topics. To evaluate iTAG, we will recruit 20 young people, ages 18-24, with HIV (YPWH) to complete 90 days worth of intervention text messages. Before and after receiving iTAG messages, they will complete computer assessments used to measure HIV medication adherence as well as other factors believed to be influence adherence such as social support. By examining participants score from before and after receiving the intervention, and by talking with participants after they receive the intervention, we hope to understand whether iTAG is acceptable to YPWH and could potential lead to improvements in their HIV treatment adherence.

DETAILED DESCRIPTION:
The current study has three aims revolved around developing and testing an intervention, called the incentivized Text-Based Adherence Game (iTAG) which is a text message-delivered intervention to improve HIV treatment adherence among Ghanaian young people with HIV (YPWH(). It expands on a prior intervention, called TAG, which used gamification strategies to improve adherence among YPWH by incorporate economic empowerment strategies including small conditional economic incentives and a peer-led mutual savings account. The central premise guiding this work is that iTAG is a feasible, acceptable, and potentially effective way to further engage YPWH in HIV care. As one of the study aims, we intend to evaluate iTAG with a single-arm pilot trial by examining YPH (N = 20-25) over 12 weeks on outcome trends, i.e., treatment adherence (i.e., antiretroviral use, viral load) and potential mediators (e.g., financial insecurity), acceptability, and indicators of feasibility and implementation potential (e.g., SMS response rate).

The single-arm pilot trial (N = 25 YPWH) will have a 12-week intervention period with pre- and-post-intervention assessments. Survey assessments will occur using an audio-assisted computer self-interview (ACASI) completed in a private space at an HIV clinic in Ghana. A post-intervention interview will also be conducted with 8 participants. Participants will be compensated for each assessment and receive phone credits for iTAG.

Final content, format, and delivery of iTAG will be determined after a prior Development Phase. Initial content, format, and delivery will be based on TAG and are as follows. YPWH receive four types of automated and tailored SMS: adherence messages (i.e., medication and clinic appointment reminders), skill messages on topics related to adherence, and story messages (i.e., SMS related to the game's storyline). Gamification strategies include themed messages, a point/reward system, and a weekly scoreboard message. Messages will also offer linkage to social support and clinic services by triggering email alerts to research staff. In addition, participants will be given opportunities to cash-in game points for mobile money or donate incentives to a mutual savings account. Code words will be used for all HIV-related topics and participants will use pseudonyms to protect privacy.

Survey assessments will be administered by SurveyToGo, an ACASI system, on tablets. The cloud system allows for encrypted storing and transfer of de-identified data collected in Ghana to research staff in the US. Participants will complete the Session Evaluation Form and the Client Satisfaction Questionnaire to assess intervention acceptability. Analytic data will also show text message (SMS) interactions for the purpose of assessing feasibility and engagement. Main outcomes will include (1) self-report of past 30-day ART adherence using a 3-item measure and (2) viral load (log10). Staff will abstract medical chart data and if viral load was not measured in the past 3 months (pre-intervention) or 1 month (post-intervention), it will be assessed at this visit as part of routine care. Secondary outcomes will also be assessed including relevant knowledge (e.g., HIV knowledge), beliefs/attitudes (e.g., attitudes towards ART), and behavior (e.g., treatment self-efficacy), social support, access to services/resources and economic wellbeing (e.g., food insecurity). A 15-min interview will also be conducted with 8 participants to further examine iTAG's acceptability and implementation potential.

Intervention acceptability will be determined using the criteria of mean scores ≥ 24 on the CSQ and ≥30 on the SEF defined as acceptable. An SMS/voice message response/receipt rate of 80% will be deemed as acceptable. To examine outcome trends, we have the following hypothesis: among the YPWH enrolled, at post-intervention, YPWH will demonstrate trends towards an increase in ART adherence and decrease in viral load (log10). They will also show improvements in secondary outcomes. Pre-post intervention differences in these outcomes will be explored using a repeated measures t-test and the Cohen's d effect size

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-24
* In treatment for HIV at our recruitment site
* Read English and speak English or a language spoken by clinic staff
* On ART medication
* Own a mobile phone
* Evidence of recent ART non-adherence
* Evidence of a detectable viral load in the past 3 months

Exclusion Criteria:

* Physically or cognitively impaired
* Participation in another ART adherence intervention

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
3-item measure of antiretroviral therapy (ART) adherence | 30 days
  This 3-item self-report survey measure assesses recent ART adherence (Wilson et al., 2016).
  Wilson, I. B., Lee, Y., Michaud, J., Fowler Jr, F. J., & Rogers, W. H. (2016). Validation of a new three-item self-report measure for medication adherence. AIDS and Behavior, 20(11), 2700-2708.
HIV viral load | Viral load testing must have been performed in past 3 months for the baseline assessment and in the past month for the 3-month follow-up assessment.
  This measure is the biological assessment HIV viral load via blood draw. Consistent with prior studies, viral load will be statistically transformed (log10) to correct for skewness.

CONTACTS AND LOCATIONS:
Locations (1):
- Komfo Anokye Teaching Hospital, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: Undecided
IDP associated with this small trial may be obtained by contacting the study's the PI.